CLINICAL TRIAL: NCT00168623
Title: Randomised Trial of Vitamin A Supplementation Given With Routine Childhood Vaccines at National Immunisation Days
Brief Title: Vitamin A Supplementation With Routine Childhood Vaccines and Mortality and Morbidity
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Bandim Health Project (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 91096-2dos03; 91096-03
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2013-11-15 (Estimated); Status verified 2013-11

CONDITIONS: Mortality; Morbidity
Keywords: Vitamin A; Vaccines; Mortality; Morbidity
MeSH Terms: interventions — Vitamin A

INTERVENTIONS:
Drug: Vitamin A

SUMMARY:
Vitamin A supplementation (VAS) is important for the immune system and may interact with different childhood vaccinations. We have hypothesized that the improved survival after VAS may depend on vitamin A amplifying the non-specific immune modulation induced by vaccinations.

In the present study we used information collected in connection with a national vitamin A campaign in Guinea-Bissau during which different doses of VAS was provided together with missing doses of DTP, OPV, and measles vaccines. We aimed to study the potential interactions between VAS and vaccine type.

DETAILED DESCRIPTION:
Vitamin A supplementation (VAS) acts as an adjuvant to vaccines, and VAS has been shown to enhance both cellular and humoral immune responses in animals and in humans. Routine childhood vaccinations have recently been shown to have important non-targeted effects on mortality, i.e. effects that cannot be explained merely by the prevention of the targeted disease. We have hypothesized that the improved survival after VAS may depend not only on the prevention of vitamin A deficiency, but also on vitamin A amplifying the non-specific immune modulation induced by routine vaccinations.

In the present study we used information collected in connection with a national vitamin A campaign in Guinea-Bissau during which different doses of VAS was provided together with missing doses of DTP, OPV, and measles vaccines. We aimed to study the potential interactions between VAS and vaccine type.

ELIGIBILITY:
Inclusion Criteria:Between 6 months and 5 years and thus eligible for vitamin A and missing vaccines during national immunisation days -

Exclusion Criteria: Overt signs of vitamin A deficiency

-

Ages: 6 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6200
Dates: Start 2003-11; Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Mortality
Morbidity
Both outcomes analysed according to vaccine received and sex

CONTACTS AND LOCATIONS:
Overall Officials: Peter Aaby, DMSc, Principal Investigator — Bandim Health Project
Locations (1):
- Bandim Health Project, Apartado 861, Bissau, Guinea-Bissau